CLINICAL TRIAL: NCT07210632
Title: Window Trial of Fluorescently Labeled Nivolumab-IRDye800 (Nivo800) in High Grade Glioma (HGG)
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Eben Rosenthal (Other)
Collaborators: Vanderbilt-Ingram Cancer Center (Other)
Responsible Party: Sponsor-Investigator, Eben Rosenthal, Barry and Amy Baker Professor and Chair, Vanderbilt-Ingram Cancer Center
Organization: Vanderbilt-Ingram Cancer Center (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: VICCHN25046
Record Dates: First submitted 2025-09-29; First posted 2025-10-07 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: Brain Cancer; HGG; Glioma; High Grade Glioma; High Grade Gliomas; High Grade Glioma (III or IV); High Grade Glioma (HGG) of the Brain With BRAF Aberration
Keywords: hgg; high grade glioma
MeSH Terms: conditions — Brain Neoplasms; Glioma | interventions — Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Nivo800 (5mg) (Experimental): 5mg nivo800
  Interventions: Drug: Nivolumab-IRDye800
- Nivo800 + Nivo (50mg +190) (Experimental): 50 mg nivo800 +190 mg nivolumab
  Interventions: Drug: Nivolumab; Drug: Nivolumab-IRDye800
- Nivo800 + Nivo (100mg + 140mg) (Experimental): 100 mg nivo800 +140 mg nivolumab
  Interventions: Drug: Nivolumab; Drug: Nivolumab-IRDye800
- Nivo800 + Nivo (150mg + 90mg) (Experimental): 150 mg nivo800 +90 mg nivolumab
  Interventions: Drug: Nivolumab; Drug: Nivolumab-IRDye800
- Nivo800 + Nivo (expansion at optimal dose cohort) (Experimental): Expansion at optimal dose
  Interventions: Drug: Nivolumab; Drug: Nivolumab-IRDye800

INTERVENTIONS:
Drug: Nivolumab — Participants will receive a single infusion of nivolumab following an infusion of nivolumab-IRDye800 (nivo800), for a combined total dose of 240 mg. This dosing applies to all cohorts except Cohort 1, which is designated as the safety group. Each cohort, other than Cohort 1, will receive no more than 240 mg in total of nivolumab and nivo800 combined. Participants will then undergo planned Standard of Care (SOC) surgical resection 1 to 4 days after the infusion.
  Arms: Nivo800 + Nivo (100mg + 140mg); Nivo800 + Nivo (150mg + 90mg); Nivo800 + Nivo (50mg +190); Nivo800 + Nivo (expansion at optimal dose cohort)
Drug: Nivolumab-IRDye800 — Participants will receive an infusion of nivolumab-IRDye800 (nivo800). Nivo800 has never been assessed in patients before and therefore Cohort 1 will receive only a test dose to determine the safety (3 participants). Cohorts 2-4 will receive escalating doses of nivo800, keeping the overall dose nivolumab + nivo800 no more than 240 mg. Participants will undergo planned Standard of Care surgical resection at 1-4 days after infusion.

SUMMARY:
High-grade gliomas (HGGs) are among the most aggressive and treatment-resistant brain tumors. Immunotherapy with checkpoint inhibitors like nivolumab has shown promise, but its efficacy remains variable and poorly understood in this patient population. This clinical trial investigates a novel imaging-enabled formulation of nivolumab-IRDye800 (nivo800) which incorporates a near-infrared (NIR) fluorescent dye to enable real-time visualization of drug distribution within tumor tissue.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent
2. Age ≥ 18 years
3. Patient must have imaging of highly suspicious high grade glioma (HGG)
4. Patients for whom surgical craniotomy is planned as standard of care (SOC)
5. Adequate hematologic and end-organ function appropriate for surgical resection and anesthesia (within 30 days of infusion) WBC ≥ 2,000 (mcl) AST 9-80 (IU/L) ALT 7-110 (IU/L) BUN 6-50 (mg/dL) Creatinine 0.5-3.0 (mg/dL) Negative hepatitis B surface antigen (HBsAg) test at screening

Exclusion Criteria:

1. Patients not eligible for SOC surgical resection
2. Active or history of autoimmune disease or immune deficiency, including, but not limited to, myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, antiphospholipid antibody syndrome, Wegener granulomatosis, Sjögren syndrome, Guillain-Barré syndrome, or multiple sclerosis with the following exceptions:

   Patients with a history of autoimmune-related hypothyroidism who are on thyroid-replacement hormone are eligible for the study.

   Patients with controlled Type 1 diabetes mellitus who are on an insulin regimen are eligible for the study.

   Patients with eczema, psoriasis, lichen simplex chronicus, or vitiligo with dermatologic manifestations only (e.g., patients with psoriatic arthritis are excluded) are eligible for the study provided if all the following conditions are met:

   Rash must cover < 10% of body surface area Disease is well controlled at baseline and requires only low-potency topical corticosteroids No occurrence of acute exacerbations of the underlying condition requiring psoralen plus ultraviolet A radiation, methotrexate, retinoids, biologic agents, oral calcineurin inhibitors, or high-potency oral corticosteroids within the previous 12 months
3. History of idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonitis, or idiopathic pneumonitis, or evidence of active pneumonitis on screening chest CT scan.

   History of radiation pneumonitis in the radiation field (fibrosis) is permitted.
4. Significant cardiovascular disease (such as New York Heart Association Class II or greater cardiac disease, myocardial infarction, or cerebrovascular accident) within 3 months prior to initiation of study treatment, unstable arrhythmia, or unstable angina.
5. Severe unresolved infection within 4 weeks prior to initiation of study treatment.
6. Prior allogeneic stem cell or solid organ transplantation
7. History of severe allergic anaphylactic reactions to chimeric or humanized antibodies or fusion proteins
8. Chronic treatment with systemic immunosuppressive medication in excess of physiologic maintenance doses of corticosteroids (>10 mg/day of prednisone or equivalent) (including, but not limited to, corticosteroids, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-TNF-a agents), with the following exceptions:

   Patients who received acute, systemic immunosuppressant medication or a dose of systemic immunosuppressant medication are eligible for the study.

   Physiologic corticosteroid replacement therapy at doses ≤ 10 mg/day of prednisone or equivalent for adrenal or pituitary insufficiency and in the absence of active autoimmune disease is permitted.

   Patients with asthma that requires intermittent use of bronchodilators, inhaled steroids, or local steroid injections may participate.

   Patients using topical, ocular, intra-articular, or intranasal steroids (with minimal systemic absorption) may participate.

   Brief courses of corticosteroids for prophylaxis (e.g., contrast dye allergy) or study treatment-related standard premedication is permitted.
9. Pregnant or breastfeeding, or intention of becoming pregnant during study treatment or within 2 months after the final dose of study treatment.
10. Participants presenting with a baseline QTcF interval > than 480 milliseconds.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2030-01-01 (Estimated); Study Completion 2031-01-01 (Estimated)

PRIMARY OUTCOMES:
Determine the safety of fluorescently labeled nivolumab-IRDye800 (nivo800) as a molecular imaging agent via assessing adverse events. | From infusion to 15 days post-infusion.
  As defined by the number of Grade ≥ 2 Adverse Events (AEs) determined that are clinically significant and considered definitely or probably related to nivo800. Safety data will be summarized by grade, severity, and type.

SECONDARY OUTCOMES:
Determine the optimal dose of nivolumab-IRDye800 (nivo800) for near-infrared (NIR) fluorescence imaging in the tumor, via microscopic imaging. | From Day of Surgery Resection to 3 months
  As defined by the lowest dose of nivo800 in a total dose of 240 mg (nivolumab + nivo800 = 240 mg) that allows for successful detection of a fluorescence signal at single cell resolution on a 4mm microscopic human tissue slide imaged under a customized Leica fluorescence microscope (20x, 2x2 binning, 3 second exposure time).

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Kelly, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Undecided
We will not share individual participant data from this pilot study due to its exploratory nature and limited sample size. Pilot studies are primarily designed to assess feasibility, refine protocols, and identify potential issues before larger-scale research is conducted. Sharing individual-level data at this stage could compromise participant confidentiality and may not yield meaningful insights given the preliminary scope of the study. Additionally, the data collected may not meet the robustness or generalizability standards required for broader dissemination.